CLINICAL TRIAL: NCT02365272
Title: Pharmacokinetic/Pharmacodynamic (PK/PD) Evaluation of Amikacin in Patients With Severe Sepsis or Septic Shock Admitted at the Emergency Department(ED)
Brief Title: Pharmacokinetic/Pharmacodynamic Evaluation Amikacin in Critically Ill Patients Admitted at the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, mevr Sabrina De Winter, PharmD - KU Leuven - University of Leuven, University Hospitals Leuven, Department of Pharmaceutical and Pharmacological Sciences B-3000 Leuven, Belgium, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: University Hospitals Leuven
Record Dates: First submitted 2015-01-27; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Sepsis
Keywords: pharmacokinetics; aminoglycosides
MeSH Terms: conditions — Sepsis | interventions — Amikacin

ARMS (2):
- amikacin standard dose (Active Comparator): amikacin in a single standard dose
  Interventions: Drug: Amikacin
- amikacin dose for critical care patients (Active Comparator): amikacin in a single dose for critical care patients
  Interventions: Drug: Amikacin

INTERVENTIONS:
Drug: Amikacin — Amikacin administered in a single dose for critical care patients

SUMMARY:
The aim of the study is the evaluation of PK/PD target attainment of amikacin in ED patients with severe sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

- patients admitted at the emergency department with a diagnosis of severe sepsis or septic shock in whom amikacin is indicatied

Exclusion Criteria:

* < 18 years
* pregnancy
* burns
* amikacin treatment in the previous 2 weeks
* known allergy to aminoglycosides
* Do Not Reanimate Code ≥ 2
* Hospitalized patients with a prolonged deep venous or arterial catheder
* Continuous renal replacement, intermittent hemodialysis and death within the time of start of amikacin replacement and 1 hour later

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with amikacin PK/PD target attainment | Participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  The primary outcome of this study was evaluation of PK/PD target attainment defined as amikacin peak concentration/Minimal Inhibitory Concentration > 8 in the 15 vs.25 mg/kg amikacin group in function of 1) actual MIC of isolated pathogens 2) breakpoints of European Committe on Antimicrobial susceptibility testing (EUCAST) of Enterobacteriaceae and Pseudomonas aeruginosa

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina De Winter, PharmD, Principal Investigator — KU Leuven - University of Leuven, University Hospitals Leuven, Department of Pharmaceutical and Pharmacological Sciences B-3000 Leuven, Belgium

REFERENCES:
- [Derived] Dia N, De Winter S, Gijsen M, Desmet S, Vanbrabant P, Peetermans W, Spriet I, Dreesen E. Dose Optimization of Amikacin in the Emergency Department: A Population Pharmacokinetics Simulation Study. Ther Drug Monit. 2025 Jun 1;47(3):353-362. doi: 10.1097/FTD.0000000000001279. Epub 2024 Dec 3. PMID 40344018
- [Derived] De Winter S, van Hest R, Dreesen E, Annaert P, Wauters J, Meersseman W, Van den Eede N, Desmet S, Verelst S, Vanbrabant P, Peetermans W, Spriet I. Quantification and Explanation of the Variability of First-Dose Amikacin Concentrations in Critically Ill Patients Admitted to the Emergency Department: A Population Pharmacokinetic Analysis. Eur J Drug Metab Pharmacokinet. 2021 Sep;46(5):653-663. doi: 10.1007/s13318-021-00698-w. Epub 2021 Jul 23. PMID 34297338
- [Derived] De Winter S, Wauters J, Meersseman W, Verhaegen J, Van Wijngaerden E, Peetermans W, Annaert P, Verelst S, Spriet I. Higher versus standard amikacin single dose in emergency department patients with severe sepsis and septic shock: a randomised controlled trial. Int J Antimicrob Agents. 2018 Apr;51(4):562-570. doi: 10.1016/j.ijantimicag.2017.11.009. Epub 2017 Nov 24. PMID 29180278